CLINICAL TRIAL: NCT02688153
Title: A Randomized Comparison of the EDWARDS INTUITY Valve System anD commErcially Available Aortic Bioprostheses in Subjects uNdergoing surgiCal Aortic Valve replacEment
Brief Title: EDWARDS INTUITY Valve System CADENCE Study
Acronym: CADENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-11
Record Dates: First submitted 2015-10-14; First posted 2016-02-23 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Aortic Valve Disease; Aortic Stenosis
Keywords: Aortic Valve Replacement; Aortic Stenosis; EDWARDS INTUITY
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EDWARDS INTUITY (Active Comparator): EDWARDS INTUITY Valve System, Model 8300A
  Interventions: Device: EDWARDS INTUITY
- Stented aortic bioprostheses (Active Comparator): Stented aortic bioprostheses
  Interventions: Device: Stented aortic bioprostheses

INTERVENTIONS:
Device: EDWARDS INTUITY — To evaluate cardiac performance characteristics and adverse events rates associated with the EDWARDS INTUITY Valve in patients undergoing AVR & CABG.
  Other Names: aortic stenosis; stenosis-based insufficiency; aortic valve replacement
  Arms: EDWARDS INTUITY
Device: Stented aortic bioprostheses — In comparison to control valves available on the market.
  Other Names: aortic stenosis; stenosis-based insufficiency; aortic valve replacement
  Arms: Stented aortic bioprostheses

SUMMARY:
The study purpose is to compare the EDWARDS INTUITY valve system with commercially available stented aortic bioprostheses, in patients requiring aortic valve replacement surgery with coronary artery bypass.

DETAILED DESCRIPTION:
This is a randomized study comparing the cross-clamp time (XCT) and cardiopulmonary bypass time (CPBT) of the EDWARDS INTUITY valve system with any commercially available stented aortic bioprosthesis, in patients with logistic EuroSCORE 1 ≥ 6 undergoing elective surgical aortic valve replacement surgery with concomitant coronary bypass grafts.

Additionally, the aim is to gather sufficient data to quantify the effect size of short term patient benefit outcomes previously identified from literature and finally to explore additional healthcare resource utilization or health economic endpoints.

ELIGIBILITY:
Inclusion:

* ≥18 years of age
* aortic stenosis / mixed aortic stenosis and aortic insufficiency
* SAVR+CABG (1-4 distal anastomoses)
* Log. EuroSCORE ≥6
* NYHA Class ≥II

Exclusion (i.a.):

* pure aortic insufficiency
* pre-existing prosthetic heart valve or ring
* congenital true bicuspid / unicuspid aortic valve
* LVEF <20%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Labrousse, MD, Principal Investigator — CHU Bordeaux - Hôpital Haut-Lévèque
Locations (1):
- CHU Bordeaux, Hôpital Haut-Lévêque, Pessac, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible subjects recruited were randomized to each arm/group as 1:1 ratio at start.
  Amongst randomized arm/group, three of the subjects randomized to the Edwards INTUITY group were converted to the control group and received commercially available surgical aortic heart valves.
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve: Subject who received an Edwards INTUITY surgical aortic heart valve.
- Control Group - Commercial Surgical Aortic Heart Valve: Subject who received a commercially available surgical aortic heart valve.
Period: Overall Study
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Started | 62 | 58
Final Randomized Arm/Group | 59 | 61
Completed | 47 | 51
Not Completed | 15 | 7
Not completed — Death | 7 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Valve Explant | 1 | 0
Not completed — Conversion to Commercial Valve | 3 | 0

BASELINE CHARACTERISTICS:
Population: Three of the subjects randomized to the Edwards INTUITY group were converted to the control group and received commercially available surgical aortic heart valves.
Units Other Than Participants: Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve | Total
Number analyzed (Participants) | 59 | 61 | 120
Number analyzed (Participants) | 59 | 61 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.4 (4.2) | 80.0 (4.8) | 79.7 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 35 | 42 | 77
Region of Enrollment [Number; unit: Participants]
  Europe | 59 | 61 | 120

OUTCOME MEASURES:

1. Primary Outcome: Average Subject Time Spent on Cardiopulmonary Cross Clamp
Description: Cardiopulmonary cross clamp time is the amount of time that the patient's aorta (blood vessel) is clamped by a surgical instrument used in cardiac surgery. This allows the normal blood flow to be sent to an artificial heart and lung machine to keep it at a constant temperature and oxygen level.
Time Frame: At time of surgery, an average of 1.5 hours
Population: The outcome is reported for subjects where data is available.
Measure: Median (Full Range); unit: Minutes
Groups:
- EDWARDS INTUITY Valve System, Model 8300A: Subject who received an Edwards INTUITY surgical aortic heart valve.
Arm/Group | EDWARDS INTUITY Valve System, Model 8300A | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 58 | 61
Minutes | 77.5 [15 to 142] | 82.0 [46 to 142]
Statistical Analysis 1: Comparison: EDWARDS INTUITY Valve System, Model 8300A vs Control Group - Commercial Surgical Aortic Heart Valve; Test type: Superiority; p = 0.3660, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -4.5

2. Primary Outcome: Average Amount of Time Subject Spent on Cardiopulmonary Bypass
Description: Cardiopulmonary bypass time is the amount of time that the patient's blood circulates through an artificial heart and lung machine during cardiac surgery.
Time Frame: At time of surgery, an average of 2 hours
Population: The outcome is reported for subjects where data is available.
Measure: Median (Full Range); unit: Minutes
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Minutes | 109.0 [53 to 179] | 107.0 [63 to 175]
Statistical Analysis 1: Comparison: Edwards INTUITY Surgical Aortic Heart Valve vs Control Group - Commercial Surgical Aortic Heart Valve; Test type: Superiority; p = 0.8377, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 2

3. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Class at 2 Years.
Description: The New York Heart Association (NYHA) functional classification system relates symptoms to everyday activities and the patient's quality of life. Class I. Patients with cardiac disease but without resulting limitation of physical activity.
  Class II. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest.
  Class III. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest.
  Class IV. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Symptoms of heart failure or the anginal syndrome may be present even at rest.
Time Frame: Baseline and 2 Years
Population: The outcome is reported for subjects where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 46 | 53
Participants
  Improved | 40 | 43
  Same | 6 | 9
  Worsend | 0 | 1

4. Secondary Outcome: Subject's Average Mean Gradients (mmHg) Measurements Over Time.
Description: Mean gradient is the average flow of blood through the aortic valve measured in millimeters of mercury. Gradients are evaluated by echocardiography over time. Mean gradient values depend on the size and type of valve.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: The outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
mmHg
  30 days: number analyzed (Participants) | 46 | 50
  30 days | 10.6 (3.9) | 10.1 (3.6)
  3 months: number analyzed (Participants) | 46 | 53
  3 months | 10.7 (4.0) | 11.1 (3.9)
  6 months: number analyzed (Participants) | 44 | 50
  6 months | 11.7 (4.3) | 11.4 (4.7)
  1 year: number analyzed (Participants) | 44 | 53
  1 year | 11.2 (4.1) | 11.5 (4.4)
  2 year: number analyzed (Participants) | 43 | 50
  2 year | 10.6 (4.4) | 11.3 (4.7)

5. Secondary Outcome: Subject's Average Peak Gradients (mmHg) Measurements Over Time.
Description: Peak gradient is the maximum value measured of flow of blood through the aortic valve as measured in millimeters of mercury. Gradients are evaluated by echocardiography over time.
Time Frame: 30 days, 3 months, 6 months, 1 year, 2 year
Population: The outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
mmHg
  30 days: number analyzed (Participants) | 46 | 50
  30 days | 19.8 (7.5) | 18.4 (6.1)
  3 months: number analyzed (Participants) | 46 | 53
  3 months | 19.5 (7.0) | 20.2 (7.3)
  6 months: number analyzed (Participants) | 44 | 50
  6 months | 21.1 (7.2) | 20.6 (8.2)
  1 year: number analyzed (Participants) | 44 | 53
  1 year | 20.0 (7.6) | 20.6 (7.7)
  2 year: number analyzed (Participants) | 43 | 50
  2 year | 19.5 (7.8) | 20.4 (8.5)

6. Secondary Outcome: Subject's Effective Orifice Area (EOA) Measurement Over Time.
Description: Effective orifice area represents the cross-sectional area of the blood flow downstream of the aortic valve. Effective orifice area is evaluated by echocardiography over time.
Time Frame: 30 days, 3 months, 6 months, 1 year, 2 year
Population: The outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: centimeters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
centimeters squared
  30 days: number analyzed (Participants) | 43 | 45
  30 days | 1.7 (0.5) | 1.6 (0.4)
  3 months: number analyzed (Participants) | 41 | 48
  3 months | 1.8 (0.6) | 1.6 (0.3)
  6 months: number analyzed (Participants) | 39 | 45
  6 months | 1.7 (0.5) | 1.6 (0.4)
  1 year: number analyzed (Participants) | 40 | 52
  1 year | 1.7 (0.4) | 1.5 (0.4)
  2 year: number analyzed (Participants) | 43 | 49
  2 year | 1.7 (0.5) | 1.5 (0.4)

7. Secondary Outcome: Subject's Effective Orifice Area Index (EOAI) Measurement Over Time.
Description: Effective orifice area index represents the minimal cross-sectional area of the blood flow downstream of the aortic valve divided by the person's body surface area. Effective orifice area index is evaluated by echocardiography over time.
Time Frame: 30 days, 3 months, 6 months, 1 year, 2 year
Population: The outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: centimeters squared/meters squared
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
centimeters squared/meters squared
  30 days: number analyzed (Participants) | 46 | 52
  30 days | 1.0 (0.3) | 0.9 (0.2)
  3 months: number analyzed (Participants) | 46 | 53
  3 months | 1.0 (0.3) | 0.9 (0.2)
  6 months: number analyzed (Participants) | 45 | 53
  6 months | 0.9 (0.3) | 0.9 (0.2)
  1 year: number analyzed (Participants) | 43 | 54
  1 year | 0.9 (0.2) | 0.8 (0.2)
  2 year: number analyzed (Participants) | 45 | 49
  2 year | 0.9 (0.3) | 0.8 (0.2)

8. Secondary Outcome: Amount of Aortic Valvular Regurgitation Over Time.
Description: Aortic valvular regurgitation occurs when the aortic valve in the heart does not close tightly allowing some of the blood that was pumped out of the heart to leak back into it. Aortic valvular regurgitation is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 represents no regurgitation and 4 represents severe regurgitation.
Time Frame: 30 days, 3 months, 6 months, 1 year, 2 year
Population: The outcome is reported for subjects where data is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days: number analyzed (Participants) | 44 | 51
  30 days: 0 None | 30 | 38
  30 days: +1 Trivial/Trace | 12 | 13
  30 days: +2 Mild | 1 | 0
  30 days: +3 Moderate | 1 | 0
  30 days: +4 Severe | 0 | 0
  3 months: number analyzed (Participants) | 43 | 48
  3 months: 0 None | 30 | 41
  3 months: +1 Trivial/Trace | 11 | 7
  3 months: +2 Mild | 0 | 0
  3 months: +3 Moderate | 2 | 0
  3 months: +4 Severe | 0 | 0
  6 months: number analyzed (Participants) | 41 | 50
  6 months: 0 None | 27 | 39
  6 months: +1 Trivial/Trace | 9 | 11
  6 months: +2 Mild | 4 | 0
  6 months: +3 Moderate | 1 | 0
  6 months: +4 Severe | 0 | 0
  1 year: number analyzed (Participants) | 40 | 49
  1 year: 0 None | 30 | 40
  1 year: +1 Trivial/Trace | 8 | 8
  1 year: +2 Mild | 1 | 1
  1 year: +3 Moderate | 1 | 0
  1 year: +4 Severe | 0 | 0
  2 year: number analyzed (Participants) | 40 | 48
  2 year: 0 None | 31 | 44
  2 year: +1 Trivial/Trace | 8 | 4
  2 year: +2 Mild | 0 | 0
  2 year: +3 Moderate | 1 | 0
  2 year: +4 Severe | 0 | 0

9. Secondary Outcome: Conversion of Edwards INTUITY Surgical Aortic Valve to Control During Surgery.
Description: Subjects randomized to the Edwards INTUITY group that were converted to the control group and received commercially available surgical aortic heart valves during surgery.
Time Frame: Prior to Surgery
Population: Original number of subjects randomized to each arm/group.
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 62 | 58
Participants | 3 | 0

10. Secondary Outcome: Subjects Who Required a Thoracic Resternotomy Over Time
Description: Number of Subjects who had a surgical opening of their chest after their initial aortic heart valve surgery shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 6 | 8
  3 months | 6 | 8
  6 months | 6 | 8
  1 year | 7 | 8
  2 year | 7 | 8

11. Secondary Outcome: Subjects Who Received a Permanent Pacemaker Over Time.
Description: Number of Subjects who received a Permanent Pacemaker shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 1 | 4
  3 months | 1 | 5
  6 months | 1 | 6
  1 year | 1 | 6
  2 year | 1 | 6

12. Secondary Outcome: Subjects With a Major Paravalvular Leak (OPC) Over Time
Description: Number of subjects who experienced a Major Paravalvular Leak (OPC) shown over various time points.
  Paravalvular leak refers to blood flowing through a channel between the implanted artificial valve and the cardiac tissue as a result of inappropriate sealing.
  Paravalvular leak is evaluated by echocardiography over time. It is assessed on a scale from 0 to 4, where 0 = no leak, 1 = a trace leak, 2 = a mild leak, 3 = a moderate leak, and 4 = a severe leak. A major paravalvular leak (OPC)are any events of leak that required surgical intervention or were considered an serious adverse event.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 1 | 0
  3 months | 1 | 0
  6 months | 1 | 0
  1 year | 1 | 0
  2 year | 1 | 0

13. Secondary Outcome: Subjects Who Experienced Major Bleeding Over Time.
Description: Number of subjects who experienced Major Bleeding shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 12 | 16
  3 months | 13 | 17
  6 months | 15 | 17
  1 year | 15 | 18
  2 year | 15 | 19

14. Secondary Outcome: Subjects Who Experienced Respiratory Failure Over Time
Description: Number of subjects who experienced a Respiratory Failure shown over various time points. Respiratory failure happens when not enough oxygen passes from your lungs to your blood.
Time Frame: 30 days, 3 Months , 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 3 | 1
  3 months | 3 | 1
  6 months | 3 | 1
  1 year | 3 | 1
  2 year | 3 | 1

15. Secondary Outcome: Subjects With a Cerebral Vascular Accident or Permanent Stroke Over Time
Description: Number of subjects who experienced a Cerebral Vascular Accident or Permanent Stroke shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 0 | 0
  3 months | 0 | 1
  6 months | 0 | 2
  1 year | 1 | 2
  2 year | 1 | 2

16. Secondary Outcome: Subjects With Renal Failure Over Time
Description: Number of subjects who experienced Renal (kidney) Failure shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 2 | 1
  3 months | 2 | 1
  6 months | 2 | 1
  1 year | 2 | 1
  2 year | 2 | 1

17. Secondary Outcome: Subjects With Endocarditis Over Time
Description: Number of subjects who experienced Endocarditis shown over various time points. Endocarditis is an infection of the endocardium, which is the inner lining of your heart chambers and heart valves.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 0 | 0
  3 months | 0 | 0
  6 months | 0 | 1
  1 year | 1 | 1
  2 year | 1 | 1

18. Secondary Outcome: Subjects With a Deep Sternal Would Infection Over Time
Description: Number of subjects who experienced a Deep Sternal Wound Infection shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 0 | 0
  3 months | 1 | 0
  6 months | 1 | 0
  1 year | 1 | 0
  2 year | 1 | 0

19. Secondary Outcome: Subjects With a Myocardial Infarction Over Time
Description: Number of subjects who experienced a Myocardial Infarction shown over various time points. A Myocardial infarction, commonly known as a heart attack, occurs when blood flow decreases or stops to a part of the heart, causing damage to the heart muscle.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 2 | 0
  3 months | 2 | 1
  6 months | 3 | 1
  1 year | 3 | 1
  2 year | 3 | 1

20. Secondary Outcome: Subjects With a Thromboembolism Over Time
Description: Number of subjects who experienced a Thromboembolism shown over various time points. A thromboembolism is an obstruction of a blood vessel by a blood clot that has become dislodged from another site in the circulation.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 2 | 0
  3 months | 2 | 2
  6 months | 3 | 3
  1 year | 4 | 4
  2 year | 5 | 4

21. Secondary Outcome: Subjects With a Cardiac Tamponade Over Time
Description: Number of subjects who experienced a Cardiac Tamponade shown over various time points. Cardiac tamponade is when fluid in the pericardium (the sac around the heart) builds up and results in compression (squeezing) of the heart.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 3 | 2
  3 months | 3 | 2
  6 months | 3 | 2
  1 year | 3 | 2
  2 year | 3 | 2

22. Secondary Outcome: Subjects With a Cardiac Reoperation for Any Reason Over Time
Description: Number of subjects who experienced a Cardiac reoperation for any reason shown over various time points.
Time Frame: 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: Cumulative number of subjects with an event by each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants
  30 days | 6 | 9
  3 months | 6 | 11
  6 months | 9 | 12
  1 year | 10 | 12
  2 year | 10 | 13

23. Secondary Outcome: Subjects Who Died Intraoperatively
Description: Number of subjects who died during surgery.
Time Frame: Surgery
Population: Number of subjects who died during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | EDWARDS INTUITY Valve System, Model 8300A | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Participants | 0 | 0

24. Secondary Outcome: Subject's Average Score on the EQ-5D- Quality of Life Questionnaire Over Time
Description: The EQ-5D is a standardized questionnaire that asks subjects to rate themselves (no problems, some problems, extreme problems) on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The scale is indexed and ranges from a minimum of 0.275 and a maximum of 1.000. A lower number indicates the participants experiences more problems and a higher number indicates the participants experiences fewer problems.
Time Frame: Baseline, 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Units on a scale
  Baseline: number analyzed (Participants) | 58 | 59
  Baseline | 0.773 (0.155) | 0.723 (0.186)
  30 day: number analyzed (Participants) | 42 | 49
  30 day | 0.790 (0.180) | 0.771 (0.189)
  3 month: number analyzed (Participants) | 48 | 51
  3 month | 0.850 (0.179) | 0.808 (0.200)
  6 month: number analyzed (Participants) | 47 | 54
  6 month | 0.877 (0.136) | 0.827 (0.206)
  1 year: number analyzed (Participants) | 41 | 53
  1 year | 0.831 (0.172) | 0.803 (0.212)
  2 year: number analyzed (Participants) | 43 | 51
  2 year | 0.864 (0.160) | 0.835 (0.198)

25. Secondary Outcome: Subject's Average Score SF-12 - Quality of Life Questionnaire Over Time
Description: The Medical Outcomes Study Short-Form 12 (SF-12) - Physical Component Summary (PCS) and Mental Component Summary (MCS).
  The SF-12 questionnaire scale ranges from 100, which reflects the best health status to 0, which reflects the worse health status.
  Subject's Average Score at Baseline and at each follow-up interval until 2 year - SF-12.
Time Frame: Baseline, 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Units on a scale
  PCS -Baseline: number analyzed (Participants) | 56 | 59
  PCS -Baseline | 40.67 (7.83) | 39.47 (7.25)
  PCS -30 day: number analyzed (Participants) | 45 | 49
  PCS -30 day | 40.57 (7.88) | 41.16 (7.02)
  PCS -3 month: number analyzed (Participants) | 48 | 52
  PCS -3 month | 44.17 (8.77) | 43.73 (8.61)
  PCS -6 month: number analyzed (Participants) | 46 | 51
  PCS -6 month | 45.87 (6.96) | 46.00 (8.47)
  PCS -1 year: number analyzed (Participants) | 42 | 51
  PCS -1 year | 45.40 (8.09) | 46.01 (8.52)
  PCS -2 year: number analyzed (Participants) | 41 | 50
  PCS -2 year | 44.74 (7.92) | 44.02 (8.35)
  MCS -Baseline: number analyzed (Participants) | 57 | 59
  MCS -Baseline | 47.30 (10.49) | 44.91 (11.16)
  MCS -30 day: number analyzed (Participants) | 45 | 50
  MCS -30 day | 48.01 (10.63) | 44.85 (11.92)
  MCS -3 month: number analyzed (Participants) | 48 | 52
  MCS -3 month | 49.56 (10.03) | 48.93 (9.46)
  MCS -6 month: number analyzed (Participants) | 46 | 51
  MCS -6 month | 50.64 (9.71) | 48.45 (10.10)
  MCS -1 year: number analyzed (Participants) | 42 | 51
  MCS -1 year | 51.08 (9.38) | 49.52 (10.09)
  MCS -2 year: number analyzed (Participants) | 41 | 50
  MCS -2 year | 51.65 (9.97) | 50.62 (9.64)

26. Secondary Outcome: Subject's Average Score on the KCCQ - Quality of Life Questionnaire Over Time
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores range from 0-100, in which higher scores reflect better health status. Subjects took this questionnaire at baseline, 30 days, 3 Months, 6 Months, 1 Year, and 2 Years.
Time Frame: Baseline, 30 days, 3 Months, 6 Months, 1 Year, 2 Years.
Population: The outcome is reported where data is available.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Units on a scale
  Baseline: number analyzed (Participants) | 58 | 59
  Baseline | 64.50 (21.95) | 57.50 (20.98)
  30 day: number analyzed (Participants) | 46 | 53
  30 day | 71.44 (22.69) | 69.24 (21.83)
  3 month: number analyzed (Participants) | 48 | 53
  3 month | 83.20 (16.26) | 78.26 (20.20)
  6 month: number analyzed (Participants) | 47 | 54
  6 month | 85.05 (15.71) | 78.74 (21.33)
  1 year: number analyzed (Participants) | 42 | 54
  1 year | 82.81 (14.86) | 80.26 (21.28)
  2 year: number analyzed (Participants) | 45 | 53
  2 year | 83.12 (18.62) | 79.31 (20.33)

27. Secondary Outcome: Health Care Utilization
Description: The average amount of time the subjects spent in the intensive care unit, the intermediate care length of stay, and the average total length of hospital stay after their heart valve replacement procedure.
Time Frame: Day of surgical procedure through discharge from the hospital, an average of 2 weeks
Population: This outcome is reported for subjects where data is available.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
Number analyzed (Participants) | 59 | 61
Days
  Length of stay | 12.0 (7.2) | 10.5 (5.3)
  ICU Length of stay: number analyzed (Participants) | 54 | 57
  ICU Length of stay | 3.9 (4.2) | 2.9 (1.9)
  Intermediate care length of stay: number analyzed (Participants) | 54 | 57
  Intermediate care length of stay | 1.2 (1.9) | 1.2 (1.4)

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through two years post implant
Groups:
- Edwards INTUITY Surgical Aortic Heart Valve: Subject who receive an Edwards INTUITY surgical aortic heart valve.
Arm/Group | Edwards INTUITY Surgical Aortic Heart Valve | Control Group - Commercial Surgical Aortic Heart Valve
All-Cause Mortality (participants affected / at risk) | 7/59 | 5/61
Serious Adverse Events (participants affected / at risk) | 42/59 | 38/61
Other Adverse Events (participants affected / at risk) | 46/59 | 43/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards INTUITY Surgical Aortic Heart Valve (N=59) | Control Group - Commercial Surgical Aortic Heart Valve (N=61)
Bleeding - cardiovascular - Major (Blood and lymphatic system disorders) | 5 | 9
Bleeding - Neurological - Major (e.g. CVA) (Blood and lymphatic system disorders) | 0 | 2
ANEMIA - BLEEDING RELATED - MINOR (Blood and lymphatic system disorders) | 1 | 1
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 1 | 1
BLOOD SEPSIS (Blood and lymphatic system disorders) | 2 | 0
BLEEDING - MUSCULOSKELETAL/DERMATOLOGICAL -MAJOR (E.G. ECCHYMOSIS) (Blood and lymphatic system disorders) | 0 | 1
BLEEDING - PERIPHERAL VASCULAR - MINOR (E.G. NOSEBLEEDS; HEMATOMAS) (Blood and lymphatic system disorders) | 0 | 1
BLEEDING - PERIPHERAL VASCULAR -MAJOR (E.G. NOSEBLEEDS; HEMATOMAS) (Blood and lymphatic system disorders) | 1 | 0
BLEEDING - GASTROINTESTINAL UPPER -MAJOR (Blood and lymphatic system disorders) | 1 | 0
BLEEDING - NEUROLOGICAL - MINOR (E.G. CVA) (Blood and lymphatic system disorders) | 1 | 0
THROMBOEMBOLIC EVENT - STROKE (Cardiac disorders) | 1 | 1
THROMBOCYTOPENIA - HEPARIN INDUCED (HIT) (Blood and lymphatic system disorders) | 1 | 0
THROMBOEMBOLIC EVENT - OTHER - PERIPHERAL - NO PARESIS (Cardiac disorders) | 1 | 0
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 3 | 4
ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 1 | 0
ARRHYTHMIA - AV BLOCK - 3RD DEGREE (Cardiac disorders) | 1 | 4
ARRHYTHMIA - BRADYCARDIA (Cardiac disorders) | 1 | 1
ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT (Cardiac disorders) | 0 | 1
ARRHYTHMIA - PERSISTANT ATRIAL FIBRILLAITON (Cardiac disorders) | 2 | 1
ARRHYTHMIA - PERMANENT ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ARRHYTHMIA - TACHYCARDIA - VENTRICULAR (Cardiac disorders) | 1 | 0
ANGINA, STABLE (Cardiac disorders) | 0 | 2
ANGINA, UNSTABLE (Cardiac disorders) | 2 | 2
CARDIAC DECOMPENSATION (Cardiac disorders) | 5 | 1
CARDIAC ARREST (Cardiac disorders) | 2 | 0
CARDIOVASCULAR - OTHER (Cardiac disorders) | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
HEART FAILURE - ACUTE (Cardiac disorders) | 1 | 2
HEART FAILURE - CHRONIC (CHF) (Cardiac disorders) | 1 | 1
CORONARY ARTERY OSTIAL OBSTRUCTION (Cardiac disorders) | 0 | 1
ENDOCARDITIS (Cardiac disorders) | 1 | 1
HYPOTENSION (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
PERICARDIAL EFFUSION - MAJOR (Cardiac disorders) | 1 | 0
HYPERTENSION - SYSTEMIC (Cardiac disorders) | 0 | 2
PERICARDIAL TAMPONADE - MAJOR (Cardiac disorders) | 2 | 0
REGURGITATION - AORTIC-CENTRAL/TRANSVALVULAR-+4 (Cardiac disorders) | 1 | 0
NSD - PARAVALVULAR LEAK - +2 (General disorders) | 1 | 0
GASTROINTESTINAL - INFECTION (Gastrointestinal disorders) | 0 | 2
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 3 | 4
RENAL FAILURE - ACUTE (Renal and urinary disorders) | 3 | 2
RENAL DYSFUNCTION (Renal and urinary disorders) | 0 | 1
GENITOURINARY - OTHER (Renal and urinary disorders) | 0 | 1
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 0 | 1
MUSCULAR SKELETAL / DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 5 | 3
BONE FRACTURE/BREAK (Musculoskeletal and connective tissue disorders) | 3 | 2
STERNAL WOUND/THORACIC INFECTION (Musculoskeletal and connective tissue disorders) | 1 | 0
NONSPECIFIC, UNKNOWN, OR OTHER BODY SYSTEM - OTHER COMPLICATION (General disorders) | 3 | 6
CANCER - NEWLY DIAGNOSED (General disorders) | 1 | 1
ANAPHYLACTIC REACTION (General disorders) | 0 | 1
MULTI-SYSTEM ORGAN FAILURE (General disorders) | 0 | 1
VASCULAR - OTHER (Vascular disorders) | 2 | 2
PLEURAL EFFUSION - LEFT (Respiratory, thoracic and mediastinal disorders) | 5 | 2
RESPIRATORY INFECTION - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
HYPOXEMIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION - RIGHT (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE -OTHER (Respiratory, thoracic and mediastinal disorders) | 2 | 1
RESPIRATORY FAILURE -ACUTE RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY DYSFUNCTION/INSUFFICIENCY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE -COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edwards INTUITY Surgical Aortic Heart Valve (N=59) | Control Group - Commercial Surgical Aortic Heart Valve (N=61)
ANEMIA - NON-BLEEDING RELATED (Blood and lymphatic system disorders) | 10 | 7
ANEMIA - BLEEDING RELATED - MINOR (Blood and lymphatic system disorders) | 6 | 0
BLEEDING - CARDIOVASCULAR - MINOR (Blood and lymphatic system disorders) | 5 | 4
ARRHYTHMIA - PAROXYSMAL ATRIAL FIBRILLATION (PAF) (Cardiac disorders) | 14 | 14
ARRHYTHMIA - AV BLOCK - 1ST DEGREE (Cardiac disorders) | 0 | 7
ARRHYTHMIA - BUNDLE BRANCH BLOCK - LEFT (Cardiac disorders) | 5 | 0
ARRHYTHMIA - BUNDLE BRANCH BLOCK - RIGHT (Cardiac disorders) | 4 | 0
ARRHYTHMIA - PERSISTANT ATRIAL FIBRILLAITON (Cardiac disorders) | 3 | 6
HYPOTENSION (Cardiac disorders) | 5 | 0
PERICARDIAL EFFUSION - MINOR (Cardiac disorders) | 4 | 0
CARDIOVASCULAR - OTHER (Cardiac disorders) | 0 | 4
URINARY TRACT INFECTION (UTI) (Renal and urinary disorders) | 7 | 9
RENAL DYSFUNCTION (Renal and urinary disorders) | 5 | 0
PSYCHIATRIC DISORDER (Psychiatric disorders) | 3 | 0
MUSCULAR SKELETAL / DERMATOLOGIC - OTHER (Musculoskeletal and connective tissue disorders) | 0 | 5
RESPIRATORY INFECTION - PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RESPIRATORY INFECTION - UPPER (URI) (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can't publish/present on overall study results not yet published but may publish his own data subject to EW review prior to submission/presentation, but data analyses of site-specific results can occur only in intervals as specified in the CTA. Publication/presentation of the PI's site-specific results of devices which haven't been market released and which still may be undergoing development, shall not include claims of device safety/effectiveness and will require the review/approval of EW.